CLINICAL TRIAL: NCT05341076
Title: Labor Scale Versus WHO Partograph for Management of Spontaneous Labor in Primigravidae (ScaLP): A Randomized Controlled Trial
Brief Title: Labor Scale Versus WHO Partograph for Management of Labor (ScaLP)
Acronym: ScaLP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sherif Abdelkarim Mohammed Shazly, M.B.B.Ch, M.S.c, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCOG1-22
Record Dates: First submitted 2022-04-11; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Dystocia
Keywords: Labor scale; Partograph; Spontaneous labor; Primigravida
MeSH Terms: conditions — Dystocia | interventions — Amniotomy; Oxytocin; Cesarean Section

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Labor scale (Experimental): Observation Amniotomy Oxytocin Cesarean Section (CS)
  Interventions: Procedure: Amniotomy; Drug: Oxytocin; Procedure: Cesarean Section
- WHO partograph (Active Comparator): Observation Amniotomy Oxytocin Cesarean Section (CS)
  Interventions: Procedure: Amniotomy; Drug: Oxytocin; Procedure: Cesarean Section

INTERVENTIONS:
Procedure: Amniotomy — Amniotomy, artificial rupture of membranes, is done with an initial delay of labor (in partograph: extension beyond the alert line, in labor scale: when progress reaches the membrane line)
  Other Names: Artificial rupture of membranes
Drug: Oxytocin — oxytocin augmentation: given with further delay of labor (according to the point of intervention of the partograph or the scale)
  Other Names: augmentation of labor
Procedure: Cesarean Section — Cesarean section: done when progress is deemed arrested (according to the definition of the partograph or the scale)
  Other Names: CS

SUMMARY:
The current study aims at evaluating the impact of the implementation of the labor scale, in comparison to the standard WHO partograph, in the management of primiparous women, including CD rate, maternal and neonatal outcomes of labor.

DETAILED DESCRIPTION:
Since the procedure was first introduced to clinical practice, Cesarean delivery (CD) has significantly contributed to peripartum maternal and fetal safety when appropriately indicated. Nevertheless, CD rate has significantly increased over the last two decades without parallel improvement in maternal or neonatal outcomes. Globally, one out of three pregnancies would be delivered by CD, resulting in growing surgical, obstetric and financial burden. Over years, long-term sequelae of current CD rate have become evident such as increased incidence of placenta accreta spectrum and exponential rise in CD trend, since 90% of women who had CD are susceptible to CD in future pregnancies. These concerns have triggered a global act to control CD rates within the margins of safe obstetric practice.

The most common indication of CD is labor dystocia. However, the definition of labor dystocia is inconsistent, and standardization of diagnosis has been heavily investigated. The WHO partograph was established at the end of the last century to serve as a tool to recognize labor dystocia and has been universally accepted to verify CD decision However, a cochrane review by Lavender et al. revealed that role of WHO partograph, in improving clinical outcomes, is lacking. In addition, there is no evidence that any published modification of the current partograph is superior to another. The "labor scale," a novel alternative to the classic partograph, was first introduced to literature in 2014. The tool was designed based on evidence-based guidelines and integrates both diagnosis and interventions to manage labor dystocia. Initial data showed that labor scale contributed to decreased incidence of CD and oxytocin administration. However, further studies are required to verify these results.

ELIGIBILITY:
Inclusion Criteria Pregnant women aged 18 to 45 years old with the following criteria: nulliparous, had been pregnant for 37 to 41 weeks with a singleton viable fetus, and vertex presented, and with estimated fetal weights between 2,500 and 4,500 g.

Exclusion Criteria Women with following criteria will be excluded: significant maternal medical or surgical comorbidity, previous uterine scar

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — N/A (study targets pregnant women in labor)
Enrollment: 206 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Successful vaginal delivery (reporting of whether labor ends in vaginal delivery or Cesarean Section. In case of CS, the indication will be reported) | Duration of labor (maximum 24 hours from onset of labor)
  The proportion who delivered vaginal versus those indicated for Cesarean Section for labor dystocia

SECONDARY OUTCOMES:
Intrapartum maternal birth injuries | Duration of labour and hospital stay (anticipated duration: 72 hours)
  This is assessed clinically at the time of labor, and includes the extent of vaginal and perineal traumas and type of repair
Primary postpartum hemorrhage | Within 24 hours of delivery
  Primary postpartum hemorrhage is defined as estimated blood loss > 500 ml following delivery and within 24 hours postpartum
Maternal fever/postpartum infections | Within 24 hours of delivery
  This is indicated by a single temperature at or above 38.0 c or 2 measurements at or above 37.5 c.
Intrapartum fetal distress | Duration of labor (maximum 24 hours)
  This criterion is met if cardiotocography shows signs consistent with pathological tracing as defined by NICE guidelines (persistent late or variable decelerations, prolonged bradaycardia or sinusoidal rhythm)
Birth injuries of the newborn | The length of neonatal hospital stay (anticipated duration: 72 hours)
  Presence of bony fractures, cephalhematoma, or intracranial hemorrhage as evident by physical examination of the newborn
Neonatal distress "asphyxia" | The length of stay in hospital/neonatal intensive care unit (anticipated duration: 72 hours)
  This is indicated by 1 and 5 minutes APGAR score, resuscitation event, umbilical artery pH, admission to neonatal intensive care unit, length of stay and any further medical complications
Duration of labor in hours | Duration of labor (maximum 24 hours)
  This starts from the onset of active labor (3 cm or more of cervical dilation) till actual delivery
Incidence of oxytocin use | Duration of labor (maximum duration: 24 hours)
  Incidence of administration of intravenous oxytocin during labor for labor augmentation
Incidence of instrumental delivery | Duration of labor (maximum duration: 24 hours)
  Instrumental delivery includes forceps and ventouse deliveries

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan Faculty of Medicine, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists (College); Society for Maternal-Fetal Medicine; Caughey AB, Cahill AG, Guise JM, Rouse DJ. Safe prevention of the primary cesarean delivery. Am J Obstet Gynecol. 2014 Mar;210(3):179-93. doi: 10.1016/j.ajog.2014.01.026. PMID 24565430
- [Background] Hamilton BE, Hoyert DL, Martin JA, Strobino DM, Guyer B. Annual summary of vital statistics: 2010-2011. Pediatrics. 2013 Mar;131(3):548-58. doi: 10.1542/peds.2012-3769. Epub 2013 Feb 11. PMID 23400611
- [Background] Gregory KD, Jackson S, Korst L, Fridman M. Cesarean versus vaginal delivery: whose risks? Whose benefits? Am J Perinatol. 2012 Jan;29(1):7-18. doi: 10.1055/s-0031-1285829. Epub 2011 Aug 10. PMID 21833896
- [Background] Neal JL, Ryan SL, Lowe NK, Schorn MN, Buxton M, Holley SL, Wilson-Liverman AM. Labor Dystocia: Uses of Related Nomenclature. J Midwifery Womens Health. 2015 Sep-Oct;60(5):485-98. doi: 10.1111/jmwh.12355. PMID 26461188
- [Background] HealthyPeople.gov. Search the Data | Healthy People 2020 [Internet]. 2017 [cited 2022 Mar 28]. p. 1-6. Available from: https://www.healthypeople.gov/2020/data-search/Search-the-Data#objid=4660;
- [Background] Tolba SM, Ali SS, Mohammed AM, Michael AK, Abbas AM, Nassr AA, Shazly SA. Management of Spontaneous Labor in Primigravidae: Labor Scale versus WHO Partograph (SLiP Trial) Randomized Controlled Trial. Am J Perinatol. 2018 Jan;35(1):48-54. doi: 10.1055/s-0037-1605575. Epub 2017 Aug 8. PMID 28787749
- [Background] Shazly SA, Embaby LH, Ali SS. The labour scale--assessment of the validity of a novel labour chart: a pilot study. Aust N Z J Obstet Gynaecol. 2014 Aug;54(4):322-6. doi: 10.1111/ajo.12209. Epub 2014 May 17. PMID 24835694
- [Background] Lavender T, Cuthbert A, Smyth RM. Effect of partograph use on outcomes for women in spontaneous labour at term and their babies. Cochrane Database Syst Rev. 2018 Aug 6;8(8):CD005461. doi: 10.1002/14651858.CD005461.pub5. PMID 30080256